CLINICAL TRIAL: NCT01963091
Title: Effect of Oxytocin on Stress Response in Cocaine-dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Megan Moran-Santa Maria, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00009981
Record Dates: First submitted 2011-07-13; First posted 2013-10-16 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxytocin (Experimental)
  Interventions: Drug: oxytocin
- placebo (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: oxytocin — Subjects will be administered 40 IUs of oxytocin nasal spray or matching placebo at 1:15pm. This dose and timing of administration was selected based on previous studies that have used similar doses of oxytocin (Ditzen, et al., 2009; Heinrichs, et al., 2003). Intranasal oxytocin and matching placebo will be compounded by Pitt Street Pharmacy Custom Compounding (Mt. Pleasant, South Carolina). Randomization will be done by a licensed pharmacist who will keep a record of the blind and be available should unblinding be necessary.
  Other Names: pitocin
  Arms: oxytocin
Drug: saline — Subjects will be administered 40 IUs of oxytocin nasal spray or matching placebo at 1:15pm. This dose and timing of administration was selected based on previous studies that have used similar doses of oxytocin (Ditzen, et al., 2009; Heinrichs, et al., 2003). Intranasal oxytocin and matching placebo will be compounded by Pitt Street Pharmacy Custom Compounding (Mt. Pleasant, South Carolina). Randomization will be done by a licensed pharmacist who will keep a record of the blind and be available should unblinding be necessary.
  Arms: placebo

SUMMARY:
Stress is associated with drug craving and relapse in substance-dependent individuals. Hormones released from the brain may mediate the behavioral response to stress. For example, several studies have indicated that oxytocin reduces stress in laboratory stress paradigms. Specifically, it appears that oxytocin promotes trust, social interaction, and calmness; yet, little is known about the potential affects of oxytocin in cocaine-dependent individuals. Given these properties of oxytocin, it may have a therapeutic role in ameliorating the negative affect commonly observed prior to relapse in cocaine-dependent individuals, as well as the anxiety associated with withdrawal. This pilot protocol will provide important preliminary data on the effect of oxytocin on stress in cocaine-dependent individuals.

ELIGIBILITY:
1) General Inclusion / Exclusion Criteria Inclusion Criteria

1. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) for a three-day period immediately prior to the CTRC admission. Nicotine dependence can affect HPA function therefore it would be ideal to exclude subjects with nicotine use. Because of the high comorbidity of cocaine and nicotine dependence, this would seriously compromise the feasibility of recruitment. In addition, because of the high comorbidity of alcohol use and cocaine dependence, individuals with alcohol abuse and dependence will be included if they do not require medically supervised detoxification. Due to the high comorbidity of cocaine and marijuana dependence, individuals with marijuana dependence will be included.
3. Subjects must consent to random assignment.
4. Subjects must consent to outpatient admission to the CTRC.

Exclusion Criteria

1. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
2. Women with premenstrual dysphoric disorder as this may impact on the response to the stress test procedure.
3. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect physiological/subjective responses.
4. Subjects with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect hormonal/neuroendocrine status.
5. Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with subjective measurements.
6. Subjects with current major depressive disorder or post-traumatic stress disorder as these disorders are associated with characteristic changes in stress response.
7. Subjects receiving synthetic glucocorticoid therapy, any exogenous steroid therapy, or treatment with other agents that interfere with hormonal measurements within one month of test session.
8. Subjects taking any psychotropic medications, opiates or opiate antagonists because these may affect test response. Subjects who have been maintained on SSRI's for 8 weeks will not be excluded.
9. Subjects with any acute illness or fever. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
10. Subjects who are > 30% over ideal weight or have a BMI greater than 35 will be considered for study participation based on the clinical judgment of study staff.
11. Subjects who are unwilling or unable to maintain abstinence from alcohol and other drugs of abuse (except nicotine) for three days prior to the stress task procedure.
12. Subjects meeting DSM-IV criteria for substance dependence (other than alcohol, nicotine, marijuana orcocaine) within the past 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Moran-Santa Maria, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Clinical Neurosciences Division-MUSC, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Salivary Cortisol Levels
Description: salivary cortisol
Time Frame: 0 minutes post 15 minute stress task
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 17 | 16
mg/dl | 0.18 (0.09) | 0.22 (0.09)

2. Secondary Outcome: Likert Scale Rating of Subjective Stress
Description: Subjects will rate subjective stress on 10-point Likert scale with 0 being 'not at all' and 10 being 'extremely'
Time Frame: 0 minutes post 15 minute stress task
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 17 | 16
units on a scale | 4.18 (3.49) | 4.25 (2.93)

3. Secondary Outcome: Likert Scale Rating of Subjective Craving
Description: Subjects will rate craving on 10-point Likert scale before and after drug administration and stress task with 0 being 'not at all' and 10 being 'extremely'
Time Frame: 0 mintues post 15 minute stress task
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 17 | 16
units on a scale | 3.35 (4.03) | 3.13 (2.80)

ADVERSE EVENTS:
Arm/Group | Oxytocin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No